CLINICAL TRIAL: NCT03772860
Title: Defining the Sympathetic Skin Response of Migraineurs in the Facial Area During the Interictal State: Comparison of Migraine Patients Who Suffer Dominant Left/Right/Bilateral Pain.
Brief Title: Defining the Sympathetic Skin Response of Migraineurs in the Facial Area
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-113-18
Record Dates: First submitted 2018-12-05; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Photic Stimulation; Acoustic Stimulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy volunteers: Healthy volunteers will be exposed to pain stimulation, visual stimulation, auditory stimulation and mental stress
  Interventions: Other: Pain stimulation; Other: Visual stimulation; Other: Auditory stimulation; Other: Mental stress
- Left headache: Migraine patients with mostly left sided headache will be exposed to pain stimulation, visual stimulation, auditory stimulation and mental stress
  Interventions: Other: Pain stimulation; Other: Visual stimulation; Other: Auditory stimulation; Other: Mental stress
- Right headache: Migraine patients with mostly right sided headache will be exposed to pain stimulation, visual stimulation, auditory stimulation and mental stress
  Interventions: Other: Pain stimulation; Other: Visual stimulation; Other: Auditory stimulation; Other: Mental stress
- Bilateral headache: Migraine patients without a dominant side headache will be exposed to pain stimulation, visual stimulation, auditory stimulation and mental stress
  Interventions: Other: Pain stimulation; Other: Visual stimulation; Other: Auditory stimulation; Other: Mental stress

INTERVENTIONS:
Other: Pain stimulation — Pain will be simulated with an electric shock 25 mlAMP over the median nerve
Other: Visual stimulation — Visual stimulation will be performed by a flicker of light on a computer screen at 15 Hrz for 0.3 seconds
Other: Auditory stimulation — Auditory stimulation will be delivered through headphones with a sound at 500 Hrz at 85 decibels for 0.3 seconds
Other: Mental stress — A mathematical challenge will be displayed on a computer screen that must be quickly solved

SUMMARY:
The aim of this study is to define the sympathetic skin response of migraineurs in the facial area. This will be achieved by exposing healthy volunteers and migraine patients to various stress stimuli (pain, visual stimulation, auditory stimulation and a mathematical challenge), and recording sympathetic skin response in the facial area.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with no history of any kind of recurrent headache
* Migraine patients according to ICH3 criteria
* Migraine patients with more than 1 attack per month

Exclusion Criteria:

* Patients with other heart or neurologic diseases
* Patients with hearing or visual decline
* Patients taking medication that effects the sympathetic system (except those taking beta blockers for migraine treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering migraine attending our Neurology Clinic and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Defining sympathetic skin response in migraineurs | One year
  Outcome will be presented as mean sympathetic response values for all the different stimuli and then separately for each stimuli

SECONDARY OUTCOMES:
Defining differences between sympathetic skin response in migraineurs | One year
  Outcome will be presented as mean sympathetic response values for all the different stimuli and then separately for each stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Yaron River, MD, Study Director — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No